CLINICAL TRIAL: NCT05707793
Title: Ultrasound Imaging of Core Muscles Activity in Multiparous Women With Vaginal Laxity: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Deraya University (Other); Minia University (Other)
Responsible Party: Principal Investigator, Doaa A. Osman, Assistant Professor, Cairo University
Other Study IDs: P.T.REC/012/004230
Record Dates: First submitted 2023-01-18; First posted 2023-02-01 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Vaginal Laxity
Keywords: ultrasound imaging; core muscles activity; multiparous women; vaginal laxity
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women suffering from vaginal laxity: self-reported perception of vaginal laxity on the Vaginal Laxity Questionnaire
  Interventions: Other: Evaluating sexual function, quality of life and pelvic floor muscle strength, as well as thickness and force (strength) of voluntary contractions of the core muscles
- normal subjects without vaginal laxity: No self-reported perception of vaginal laxity on the Vaginal Laxity Questionnaire
  Interventions: Other: Evaluating sexual function, quality of life and pelvic floor muscle strength, as well as thickness and force (strength) of voluntary contractions of the core muscles

INTERVENTIONS:
Other: Evaluating sexual function, quality of life and pelvic floor muscle strength, as well as thickness and force (strength) of voluntary contractions of the core muscles — Evaluation through Vaginal Laxity Questionnaire, Female Sexual Function Index, Short-Form 36 Health Survey, modified Oxford grading scale and ultrasound imaging

SUMMARY:
This study aims to compare the ultrasound imaging of core muscles activity in multiparous women with vaginal laxity versus normal controls.

DETAILED DESCRIPTION:
Vaginal laxity is characterized by the loss of elasticity in the vaginal structure and vaginal looseness, which leads to symptoms including sexual dysfunction, dyspareunia, chronic pelvic pain, and urinary incontinence. It is a symptom of pelvic floor dysfunction. Its mechanisms are not well understood and it is usually worse in women with multiparity.

Since the pelvic floor muscles (PFMs) are one of the core muscles that play a critical role in lumbopelvic stability, their impairment may affect the lumbopelvic area and the activity of other core muscles, like the transverse abdominis, lumbar multifidus, and diaphragm. Therefore, this study aims to compare the ultrasound imaging of core muscles activity in multiparous women with vaginal laxity versus normal controls.

ELIGIBILITY:
Inclusion Criteria:

1. The participants' age range from 35 to 45 years
2. their body mass index is 25-30 kg/m2,
3. The number of normal deliveries ≤ three times,
4. having a regular menstruation.
5. They participate in the study after at least two years from their last delivery.

Exclusion Criteria:

1. Prior history of disc prolapse and sacroiliac joints, symphysis pubic joint as well as lower limb problems, leg length discrepancy, and diastasis recti.
2. Surgery related to the spine, abdomen or pelvis.
3. Genital prolapse, urinary tract infection, and intrauterine device.
4. Diabetes, chest and/or cardiac disease.
5. Using any drugs for sexual dysfunction.

Ages: 35 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: referred by gynecologists from the outpatient clinic for gynecology, Minia university Hospital, Minia, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
ِAssessment of diaphragmatic force | 3 months
  Diaphragmatic excursion will be measured, using an ultrasound device, by placing calipers at the bottom and top of the diaphragmatic inspiratory slope. All measurements will be taken at the end of expiration phase for women in both groups.
Assessment of transverse abdominis thickness | 3 months
  The measurement of transverse abdominis muscle will be taken from the lower border of internal obliques muscle to the inferior hyperechoic line of peritoneum at rest and during the abdominal drawing in maneuvers (ADIM) for women in both groups, using an ultrasound device.
Assessment of lumbar multifidus thickness | 3 months
  Lumbar multifidus will be measured, using an ultrasound device, along the line from the L4-5 zygapophyseal joint to the superior border of the lumbar multifidus for women in both groups.
Assessment of pelvic floor muscle force | 3 months
  It will be assessed, using an ultrasound device, for women in both groups. The position of the bladder base at rest will be marked electronically with an 'X'. The subject will then perform a maximum voluntary pelvic floor muscle contraction and the image will be captured at the moment of maximum displacement. At this time, the subject will relax the pelvic floor muscles. The investigator will then measure the displacement to its current position in the stilled image and will be blinded to the measurement value until after the caliper has been fixed at the end point.

SECONDARY OUTCOMES:
Vaginal Laxity Questionnaire | 3 months
  It is the only available tool for vaginal laxity assessment. Therefore, it will be used to exclude the diagnosis of vaginal laxity for women in group (A) and to confirm the diagnosis of vaginal laxity for women in group (B) through asking women to score vaginal laxity on a scale of 1 to 7, with 1 being very loose and 7 being very tight (Krychman et al., 2017).
The Female Sexual Function Index (FSFI) | 3 months
  The Female Sexual Function Index (FSFI) is a brief, multidimensional self-report instrument that will be used to assess the key dimensions of sexual function for women in both groups. The scale consists of 19 items yields domain scores in the following six areas: sexual desire, arousal, lubrication, orgasm, satisfaction and pain (Zachariou et al., 2017).
Short-Form 36 Health Survey (SF-36) | 3 months
  It will be used to assess the quality of life for women in both groups. The scale is intended to assess disease burden and to assess the patient's quality of life as an indication of the patient's health status. It consists of 36 questions that evaluate eight domains: physical functioning (the ability to care for oneself and perform daily tasks); role limitations caused by physical health problems (the impact of one's physical health on one's capacity to perform daily tasks); bodily pain (the level of pain experienced whilst performing daily tasks); general health perceptions (how one sees one's own health); vitality (the capacity to carry out daily tasks); and social functioning. Scores range from zero (most affected) to one hundred (not affected) (Ramage et al., 2017).
Modified Oxford grading scale | 3 months
  The modified Oxford grading scale (with scores from 0 to 5) will be used to evaluate the pelvic floor muscle strength for women in both groups through measuring the vaginal digital palpation in a crock-lying position (Ferreira et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Osman, Assis. Prof., Principal Investigator — Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Minia university Hospital, Minya, Minya Governorate, Egypt